CLINICAL TRIAL: NCT03612297
Title: Impact of Selective Reporting of Antibiotic Susceptibility Test Results in Urinary Tract Infections in the Outpatient Setting: a Protocol for a Pragmatic, Prospective Quasi-experimental Trial
Brief Title: Selective Reporting of Antibiotic Susceptibility Test Results in Urinary Tract Infections in the Outpatient Setting
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: PREPS-17-0026
Record Dates: First submitted 2018-07-02; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-06

CONDITIONS: Urinary Tract Infections
Keywords: Antimicrobial resistance; Antimicrobial stewardship; Selective reporting antimicrobial susceptibility tests; Escherichia coli
MeSH Terms: conditions — Urinary Tract Infections; Escherichia coli Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ATOUTBIO: Selective reporting of antibiotic susceptibility tests for all E. coli identified in urine cultures of adults.
  Interventions: Diagnostic Test: Selective reporting of Antibiotic Susceptibility Tests
- EVOLAB: Complete reporting of antibiotic susceptibility tests for all E. coli identified in urine cultures of adults.

INTERVENTIONS:
Diagnostic Test: Selective reporting of Antibiotic Susceptibility Tests — Selective reporting of antibiotic susceptibility tests for all E. coli identified in urine cultures of adults: results of susceptibility are reported back to the practitioner only for few (n=5-6) antibiotics, those that should be used in first line according to guidelines. Susceptibility results not mentioned in the selective reporting of AST are available at the practitioners' request to the microbiologist. Data used to determine which antibiotic to report for UTIs are the isolated microorganism, the patient age and gender, and antibiotics recommended in national guidelines. As guidelines for UTIs treatment differ by gender, two algorithms have been developed and pilot-tested by three GPs, one microbiologist and two infectious disease physicians.
  Groups: ATOUTBIO

SUMMARY:
Antibiotic resistance is a serious and increasing worldwide threat to global public health. One of antibiotic stewardship programmes' objectives is to reduce inappropriate broad-spectrum antibiotics' prescription. Selective reporting of antibiotic susceptibility test (AST) results, which consists of reporting to prescribers only few (n=5-6) antibiotics, preferring first-line and narrow-spectrum agents, is one possible strategy advised in recommendations. However, selective reporting of AST has never been evaluated using an experimental design.

This study is a pragmatic, prospective, multicentre, controlled (selective reporting vs usual complete reporting of AST), before-after (year 2019 vs 2017) study. Selective reporting of AST is scheduled to be implemented from September 2018 in the ATOUTBIO group of 21 laboratories for all E. coli identified in urine cultures in adult outpatients, and to be compared to the usual complete AST performed in the EVOLAB group of 20 laboratories. The main objective is to assess the impact of selective reporting of AST for E. coli positive urine cultures in the outpatient setting on the prescription of broad-spectrum antibiotics frequently used for urinary tract infections (amoxicillin-clavulanate, third generation cephalosporins and fluoroquinolones). The primary endpoint is the after (2019) - before (2017) difference in prescription rates for the previously mentioned antibiotics/classes that will be compared between the two laboratory groups, using linear regression models. Secondary objectives are to evaluate the feasibility of selective reporting of AST implementation by French laboratories and their acceptability by organising focus groups and individual semi-structured interviews with general practitioners and laboratory professionals.

DETAILED DESCRIPTION:
Antibiotic resistance (ABR) is a serious and increasing worldwide threat to global public health. It has been estimated that multidrug-resistant bacteria affect 158.000 French persons annually, of whom 12.500 die from these infections. In France, the increase of multidrug resistance among Enterobacteriaceae is the most alarming: the prevalence of Escherichia coli resistant to third generation cephalosporins and to fluoroquinolones has dramatically increased in the last decade and has reached now 11% and 17%, respectively. More than 90% of antibiotics used in humans in France are prescribed to outpatients (70% by general practitioners) and urinary tract infections (UTIs) account for a considerable proportion of these prescriptions (15% of all outpatient prescriptions, about 10 million of prescriptions each year) with E. coli being the pathogen most frequently (70-95%) isolated in community-acquired UTIs. Antibiotic stewardship programmes aim both at limiting antibiotic therapy to proven or strongly suspected non-self-limiting bacterial infections, and at reducing broad-spectrum antibiotics' use, such as amoxicillin-clavulanate, cephalosporins and fluoroquinolones. So, two goals are pursued: to avoid unnecessary antibiotic use, and to limit inappropriate antibiotic prescribing. Several studies have shown that half of antibiotic prescriptions for UTIs in primary care are either unnecessary or inappropriate, and that general practitioners (GPs) prescribe more antibiotics than necessary. Broad-spectrum antibiotics (in particular amoxicillin-clavulanate, cephalosporins and fluoroquinolones) are frequently inappropriately prescribed in UTIs, whereas first-line and narrow-spectrum antibiotics (e.g. amoxicillin, nitrofurantoin, fosfomycin, etc.) would have been sufficient to treat the infection.

One strategy recommended by French national authorities and by international recommendations to limit the inappropriate over-prescription of broad-spectrum antibiotics is the use of selective reporting for antibiotic susceptibility test (AST) results. Selective reporting means that AST are reported back to the practitioner only for few (n=5-6) antibiotics, those that should be used first-line according to guidelines. However, the laboratory is still testing all the 20-25 antibiotics reported in the usual complete AST, and susceptibility results not mentioned in the selective reporting of AST are available at the practitioners' request to the microbiologist. Data usually used to determine which antibiotics to report for urine samples are the isolated microorganism, the patient's age and gender, and the list of antibiotics recommended in national guidelines. For example, in a wild-type E. coli isolated in urine in an adult woman, the only antibiotics to report could be amoxicillin, trimethoprim/sulfamethoxazole, nitrofurantoin, fosfomycin and pivmecillinam. To date however, even if recommended by the French authorities, selective reporting of AST is still limited to rare local initiatives. Two randomised controlled case-vignette surveys conducted among junior medical doctors and GPs in France revealed that selective reporting of AST could improve the appropriateness of antibiotic treatment for UTIs and decrease the prescription of broad-spectrum antibiotics, while being well accepted by most physicians. However, these two surveys used fictitious clinical vignettes and no study has yet been conducted in the 'real life' French health context to evaluate the impact of selective reporting of AST on antibiotic prescribing.

METHODS

Study objectives

The main objective of this study is to assess the impact of selective reporting of AST for E. coli positive urine cultures in adult outpatients on the prescription of broad-spectrum antibiotics frequently used in UTIs (amoxicillin-clavulanate, third generation cephalosporins and fluoroquinolones). These antibiotics/classes have been indeed flagged since 2013 as 'critical' antibiotics (i.e. antibiotics with a higher risk of selection of bacterial resistance) by the French Medicines Agency, in line with the recent AWaRe categorisation introduced by the WHO in its Essential Medicines List. Secondary objectives are to evaluate the feasibility of the selective reporting of AST implementation by French laboratories and their acceptability by GPs and laboratory professionals (microbiologists, technicians and secretaries).

Study design and setting

This study is a pragmatic, prospective, multicentre, controlled (selective reporting vs usual complete reporting of AST), before-after study. Selective reporting of AST is scheduled to be implemented, from the 1st of September 2018, in the ATOUTBIO group of 21 laboratories for all E. coli identified in urine cultures of adults, and to be compared to the complete reporting of AST performed in the EVOLAB group of 20 laboratories. ATOUTBIO and EVOLAB are the two main laboratory networks located in Lorraine (north-eastern France region with a population of 2,346,000 according to the 2014 census), and each of them is set up on approximatively one third of the regional territory. The target study population is adults, with an E. coli positive urine culture on which an AST is realised, (according to national recommendations), who are prescribed an antibiotic by primary care physicians (GPs and other specialties) located in the geographic areas served by all the 41 laboratories studied (in the intervention ATOUTBIO group or the control EVOLAB group). The 'before' period is the year preceding the implementation of selective reporting of AST in the ATOUTBIO group (i.e. the 2017 year) and the 'after' period is the year following this implementation (i.e. the 2019 year). The feasibility of the intervention for laboratories is evaluated by collecting prospectively in a database all material/informatics, financial and human laboratory resources used in 2018 and 2019 for the implementation of selective reporting of AST. The acceptability of the intervention is assessed by organising focus groups and individual semi-structured interviews with a randomised sample of GPs and laboratory professionals to collect their perceptions on selective reporting of AST one year after its implementation (September 2019). The monthly number of complete reporting of AST requested by physicians is also calculated as an indicator of prescribers' acceptability. This study complies with existing methodology guidance for stewardship studies.

Study organisation

This study is promoted and coordinated by Nancy University Teaching Hospital. A scientific committee is in charge of supervising all scientific aspects and organisational issues occurring during the study period. This committee is multidisciplinary, comprising four microbiologists, two infectious diseases physicians, one GP, one epidemiologist and public health specialist, one sociologist and one pharmacist. The committee will meet regularly: at least one meeting before the study starts to define the protocol, at least two meetings per year during the study period to solve organizational issues, and at least one meeting after the end of the study period to present and discuss the results.

Description of the intervention: selective reporting of AST

As French guidelines for UTIs' treatment differ by gender, two algorithms have been developed and pilot-tested by three GPs, one microbiologist and two infectious diseases physicians. During the algorithms' development, two possible risks associated with selective reporting of AST have been taken into account. First, physicians may have problems prescribing an antibiotic for patients with multiple allergies or contra-indications; indeed, for each possible clinical situation, at least two different classes of antibiotics are reported on the selective report and the sentence 'the complete AST is available at the prescriber' request is specifically mentioned on the report. Second, as the clinical diagnosis is unknown to the microbiologist and then, in order to avoid the increased use of antibiotics reported on the selective report but not appropriate to the clinical context (e.g. nitrofurantoin in pyelonephritis as previously reported in other studies), antibiotics that should not be used in pyelonephritis or prostatitis are specifically flagged on the report.

Data collected

Data collected for each AST performed on E. coli positive urine cultures in 2017 (before period) and 2019 (after period) in all laboratories of the two groups are: patient's gender and age, living residence (community/nursing home), study group (intervention (ATOUTBIO)/control (EVOLAB)), antibiotic(s) dispensed by a community pharmacy during the 15 days following the AST (yes/no, molecule(s), dosage, type of package and quantity), and the prescriber's speciality. During the 'after period', the number of medical consultations and hospitalisations during the 30 days following the AST are collected, in order to look for any unintended consequences. All these data stem from the French health insurance database SNDS (Système National des Données de Santé) that contains individualised, anonymous and linkable data. Prospectively recorded for all beneficiaries of healthcare in France, SNDS covers almost the entire French population (67 million inhabitants). Data recorded include especially all medical expenditure reimbursements (all antibiotics are reimbursed in France) and information from hospital stays. The SNDS database is one of the largest databases in the world that has been extensively used to guide public health policies in France. A probabilistic data linkage method is applied within the anonymous SNDS database to identify patients for which urine cultures positive for E. coli and with an AST were processed in 2017 and 2019 in the two groups of laboratories.

Sample size

Based on national published data, the prescription rate of broad-spectrum antibiotics frequently used in UTIs is estimated to be at around 70% in French outpatients. A sample of 300 urine cultures positive for E. coli and with an AST per group would be sufficient to detect a 10% decrease difference in the prescription rate between groups after intervention, with a 90% power, a 5% α risk and an inflation factor at 3 (due to the cluster design). The two laboratory networks included in this study will definitely be sufficient to detect such a difference as more than 16,000 AST on E. coli urine cultures are performed each year by both EVOLAB and ATOUTBIO groups.

Statistical analyses

The statistical analysis plan includes the following procedures: (i) A comparison of laboratory activities between the two groups (ATOUTBIO and EVOLAB) in 2017 and 2019: number of AST in urine cultures, E. coli prevalence in urine cultures, antibiotic resistance profiles of E. coli isolated from urine cultures, (ii) A comparison of age and sex-ratio of patients with E. coli positive urine cultures (with AST) between the two groups in 2017 and 2019, (iii) The calculation, for each laboratory group, of the prescription rates in suspected UTIs of amoxicillin-clavulanate, third generation cephalosporins, fluoroquinolones and all these three antibiotics/classes combined in 2017 and 2019, as follows: number of prescriptions of antibiotic/class y for E. coli positive urine cultures with AST during the year n / number of prescriptions of all antibiotics for E. coli positive urine cultures with AST during the year n, (iv) A comparison of the after (2019) - before (2017) difference of the prescription rates for the above-mentioned antibiotics/classes between the two groups, using linear regression models adjusted for variables that might differ between groups (laboratory activities, sex-ratio, age).

A p-value of < 0.05 for two-sided tests is considered significant. All analyses are performed with SAS version 9.4 (SAS Institute, Inc., Cary, N.C.).

ELIGIBILITY:
Inclusion Criteria:

* adults with an E. coli positive urine culture on which an AST is realised in the year 2017 and 2019 in ATOUTBIO or EVOLAB laboratories
* adults who go to ambulatory care practitioners located in the geographic areas served by all the 41 laboratories studied (in the intervention ATOUTBIO group or the control EVOLAB group).

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with E. coli urinary tract infections
Sampling Method: Probability Sample
Enrollment: 64000 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Impact of selective reporting of AST for E. coli positive urine cultures in outpatient setting on the prescription of broad-spectrum antibiotics frequently used on UTIs (amoxicillin-clavulanate, third generation cephalosporins and fluoroquinolones) | 2 years (1 year before + 1 year after)
  A comparison of the after (2019) - before (2017) difference of the prescription rates for previous mentioned antibiotics/classes between the two groups, using linear regression models adjusted for variables that differ between groups (laboratory activities, sex-ratio, age).

SECONDARY OUTCOMES:
Laboratory expenditures (in euros) for the implementation of the intervention | 2 years
  Collection of all laboratory expenditures made in euros in 2018 and 2019 for the implementation of the selective reporting of AST.
Satisfaction of GPs and laboratory staffs about selective reporting of AST, assessed by a visual analog scale | 1 year
  The visual analog scale is a likert scale varying from 0 to 10. Satisfaction will be collected by organizing focus groups and individual semi-structured interviews with a randomised sample of GPs and laboratory staffs one year after the selective reporting of AST implementation (September 2019).

CONTACTS AND LOCATIONS:
Overall Officials: Céline Pulcini, Professor, Principal Investigator — Central Hospital, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Etienne C, Pulcini C. [Prospective cross-sectional study of antibiotic prescriptions in a sample of French general practitioners]. Presse Med. 2015 Mar;44(3):e59-66. doi: 10.1016/j.lpm.2014.07.022. Epub 2015 Jan 31. French. PMID 25650299
- [Background] Denes E, Prouzergue J, Ducroix-Roubertou S, Aupetit C, Weinbreck P. Antibiotic prescription by general practitioners for urinary tract infections in outpatients. Eur J Clin Microbiol Infect Dis. 2012 Nov;31(11):3079-83. doi: 10.1007/s10096-012-1668-9. Epub 2012 Jun 22. PMID 22722765
- [Background] Barlam TF, Cosgrove SE, Abbo LM, MacDougall C, Schuetz AN, Septimus EJ, Srinivasan A, Dellit TH, Falck-Ytter YT, Fishman NO, Hamilton CW, Jenkins TC, Lipsett PA, Malani PN, May LS, Moran GJ, Neuhauser MM, Newland JG, Ohl CA, Samore MH, Seo SK, Trivedi KK. Implementing an Antibiotic Stewardship Program: Guidelines by the Infectious Diseases Society of America and the Society for Healthcare Epidemiology of America. Clin Infect Dis. 2016 May 15;62(10):e51-77. doi: 10.1093/cid/ciw118. Epub 2016 Apr 13. PMID 27080992
- [Background] Pulcini C, Tebano G, Mutters NT, Tacconelli E, Cambau E, Kahlmeter G, Jarlier V; EUCIC-ESGAP-EUCAST Selective Reporting Working Group. Selective reporting of antibiotic susceptibility test results in European countries: an ESCMID cross-sectional survey. Int J Antimicrob Agents. 2017 Feb;49(2):162-166. doi: 10.1016/j.ijantimicag.2016.11.014. Epub 2017 Jan 10. PMID 28093208
- [Background] Coupat C, Pradier C, Degand N, Hofliger P, Pulcini C. Selective reporting of antibiotic susceptibility data improves the appropriateness of intended antibiotic prescriptions in urinary tract infections: a case-vignette randomised study. Eur J Clin Microbiol Infect Dis. 2013 May;32(5):627-36. doi: 10.1007/s10096-012-1786-4. Epub 2012 Dec 8. PMID 23224717
- [Background] Bourdellon L, Thilly N, Fougnot S, Pulcini C, Henard S. Impact of selective reporting of antibiotic susceptibility test results on the appropriateness of antibiotics chosen by French general practitioners in urinary tract infections: a randomised controlled case-vignette study. Int J Antimicrob Agents. 2017 Aug;50(2):258-262. doi: 10.1016/j.ijantimicag.2017.01.040. Epub 2017 May 31. PMID 28577933
- [Background] Silveira DP, Artmann E. Accuracy of probabilistic record linkage applied to health databases: systematic review. Rev Saude Publica. 2009 Oct;43(5):875-82. doi: 10.1590/s0034-89102009005000060. Epub 2009 Sep 25. English, Portuguese. PMID 19784456
- [Background] Langford BJ, Seah J, Chan A, Downing M, Johnstone J, Matukas LM. Antimicrobial Stewardship in the Microbiology Laboratory: Impact of Selective Susceptibility Reporting on Ciprofloxacin Utilization and Susceptibility of Gram-Negative Isolates to Ciprofloxacin in a Hospital Setting. J Clin Microbiol. 2016 Sep;54(9):2343-7. doi: 10.1128/JCM.00950-16. Epub 2016 Jul 6. PMID 27385708
- [Background] Steffee CH, Morrell RM, Wasilauskas BL. Clinical use of rifampicin during routine reporting of rifampicin susceptibilities: a lesson in selective reporting of antimicrobial susceptibility data. J Antimicrob Chemother. 1997 Oct;40(4):595-8. doi: 10.1093/jac/40.4.595. PMID 9372433
- [Background] Johnson LS, Patel D, King EA, Maslow JN. Impact of microbiology cascade reporting on antibiotic de-escalation in cefazolin-susceptible Gram-negative bacteremia. Eur J Clin Microbiol Infect Dis. 2016 Jul;35(7):1151-7. doi: 10.1007/s10096-016-2645-5. Epub 2016 Apr 29. PMID 27130036
- [Background] Tan TY, McNulty C, Charlett A, Nessa N, Kelly C, Beswick T. Laboratory antibiotic susceptibility reporting and antibiotic prescribing in general practice. J Antimicrob Chemother. 2003 Feb;51(2):379-84. doi: 10.1093/jac/dkg032. PMID 12562706
- [Background] McNulty CA, Lasseter GM, Charlett A, Lovering A, Howell-Jones R, Macgowan A, Thomas M. Does laboratory antibiotic susceptibility reporting influence primary care prescribing in urinary tract infection and other infections? J Antimicrob Chemother. 2011 Jun;66(6):1396-404. doi: 10.1093/jac/dkr088. Epub 2011 Mar 11. PMID 21398297
- [Background] Sharland M, Pulcini C, Harbarth S, Zeng M, Gandra S, Mathur S, Magrini N; 21st WHO Expert Committee on Selection and Use of Essential Medicines. Classifying antibiotics in the WHO Essential Medicines List for optimal use-be AWaRe. Lancet Infect Dis. 2018 Jan;18(1):18-20. doi: 10.1016/S1473-3099(17)30724-7. Epub 2017 Dec 20. No abstract available. PMID 29303731
- [Background] Pulcini C, Huttner A. CMI policy on antimicrobial stewardship research. Clin Microbiol Infect. 2018 Feb;24(2):91-92. doi: 10.1016/j.cmi.2017.11.006. Epub 2017 Nov 10. No abstract available. PMID 29133158
- [Background] Tuppin P, Rudant J, Constantinou P, Gastaldi-Menager C, Rachas A, de Roquefeuil L, Maura G, Caillol H, Tajahmady A, Coste J, Gissot C, Weill A, Fagot-Campagna A. Value of a national administrative database to guide public decisions: From the systeme national d'information interregimes de l'Assurance Maladie (SNIIRAM) to the systeme national des donnees de sante (SNDS) in France. Rev Epidemiol Sante Publique. 2017 Oct;65 Suppl 4:S149-S167. doi: 10.1016/j.respe.2017.05.004. Epub 2017 Jul 27. PMID 28756037
- See also: Santé publique France. Résistance aux anti-infectieux - Données par pathogène. 2017. — http://invs.santepubliquefrance.fr/Dossiers-thematiques/Maladies-infectieuses/Resistance-aux-anti-infectieux/Donnees-par-pathogene
- See also: Agence nationale de sécurité du médicament et des produits de santé. L'évolution des consommations d'antibiotiques en France entre 2000 et 2015 — http://ansm.sante.fr/S-informer/Points-d-information-Points-d-information/Evolution-des-consommations-d-antibiotiques-en-France-entre-2000-et-2015-Point-d-Information
- See also: Société de Pathologie Infectieuse de Langue Française. Recommandations pour la prise en charge des infections urinaires bactériennes communautaires de l'adulte. 2017. — http://infectiologie.com/fr/actualites/infections-urinaires-communautaires-maj2017_-n.html
- See also: Ministère chargé de la santé. Plan national d'alerte sur les antibiotiques. 2011-2016. — http://solidarites-sante.gouv.fr/IMG/pdf/plan_antibiotiques_2011-2016_DEFINITIF.pdf
- See also: Ministère des Solidarités et de la Santé. La mise en place d'antibiogrammes ciblés dans les infections urinaires à Escherichia coli. 2016 — http://solidarites-sante.gouv.fr/IMG/pdf/antibiogrammes_cibles_ps.pdf